CLINICAL TRIAL: NCT01878461
Title: A Randomized, Vehicle Controlled, Double Blind, Parallel Group, Multi Center PhaseIII Study to Evaluate the Safety and Efficacy of M518101 in Subjects With Plaque Psoriasis
Brief Title: Evaluate the Efficacy and Safety of M518101 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M518101-US03
Record Dates: First submitted 2013-06-06; First posted 2013-06-17 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Proper quantity twice a day
  Interventions: Drug: Vehicle
- M518101 (Experimental): Proper quantity twice a day
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: Vehicle
  Arms: Vehicle
Drug: M518101
  Arms: M518101

SUMMARY:
This study is to evaluate the efficacy and safety of M518101 in subjects with plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Who are able and willing to give signed informed consent
* Who are male or females aged 18 years or older with plaque psoriasis confirmed by the Investigator.
* Who have up to 20% of body surface area (BSA) afflicted with plaques
* Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

* Who have a history of allergy to vitamin D3 derivative preparations or a history of relevant drug hypersensitivity.
* Who are pregnant or lactating.
* Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
* Who are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
* Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study
* Whose serum calcium levels exceed the upper limit of reference range
* Who have used any investigational medicinal product and/or participated in any clinical study within 60 days of randomization.
* Who have been treated with systemic therapy within 30days of randomization.
* Who have treated with biologics within 5 half-lives of the biologics before the day of randomization
* Who have been treated with topical therapy within 14days before the day of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | 8 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Agave Clinical Research, Mesa, Arizona
  - T Joseph Raoof, Encino, California
  - Medical Center for Clinical Research, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Horizons Clinical Research Center, Denver, Colorado
  - The Center for Clinical and Cosmetic Research, Aventura, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Northshore University Health System, Skokie, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Kansas City Dermatology, Overland Park, Kansas
  - Derm Research, Louiville, Kentucky
  - Dermatology Specialists Research, Lousville, Kentucky
  - Medical Development Center, Baton Rouge, Louisiana
  - Grekin Skin Institute, Warren, Michigan
  - Washington University Dermatology, St Louis, Missouri
  - Karl G Heine Dermatology, Henderson, Nevada
  - Las Vegas Skin and Cancer Center, Las Vegas, Nevada
  - Center of Central New Jersey, East Windsor, New Jersey
  - Skin Search of Rochester, Rochester, New York
  - Derm Research Center of New York, Stony Brook, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Medical Development Center, Wilmington, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Palmetto Clinical Trial Servises, Fountain Inn, South Carolina
  - Coastal Clinical Research Center, Mt. Pleasant, South Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Austin Dermatology Associates, Austin, Texas
  - DermResearch, Austin, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah